CLINICAL TRIAL: NCT04565665
Title: Study of Cord Blood Derived Mesenchymal Stem Cells for Treatment of Moderate, Severe or Critical Pneumonia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-0365; NCI-2020-06741 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0365 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-09-22; First posted 2020-09-25 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-09

CONDITIONS: COVID-19 Infection; COVID-19-Associated Acute Respiratory Distress Syndrome; Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm; Symptomatic COVID-19 Infection Laboratory-Confirmed
MeSH Terms: conditions — COVID-19; Hematologic Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase II Arm I (mesenchymal stem cells) (Experimental): Patients receive MSCs as in the Pilot study.
  Interventions: Biological: Mesenchymal Stem Cell
- Phase II Arm II (standard of care) (Active Comparator): Patients receive standard of care.
  Interventions: Other: Best Practice
- Pilot study (mesenchymal stem cells) (Experimental): Patients receive MSCs IV over 1-2 hours on day 1. Patients may receive a second infusion of MSCs within 7 days after the first infusion per physician discretion.
  Interventions: Biological: Mesenchymal Stem Cell

INTERVENTIONS:
Other: Best Practice — Receive standard of care
  Other Names: standard of care; standard therapy
  Arms: Phase II Arm II (standard of care)
Biological: Mesenchymal Stem Cell — Given IV
  Other Names: Mesenchymal Progenitor Cell; MPC
  Arms: Phase II Arm I (mesenchymal stem cells); Pilot study (mesenchymal stem cells)

SUMMARY:
This is a phase I trial followed by a phase II randomized trial. The purpose of phase I study is the feasibility of treating patients with acute respiratory distress syndrome (ARDS) related to COVID-19 infection (COVID-19) with cord blood-derived mesenchymal stem cells (MSC). The purpose of the phase II trial is to compare the effect of MSC with standard of care in these patients. MSCs are a type of stem cells that can be taken from umbilical cord blood and grown into many different cell types that can be used to treat cancer and other diseases. The MSCs being used for infusion in this trial are collected from healthy, unrelated donors and are stored and grown in a laboratory. Giving MSC infusions may help control the symptoms of COVID-19 related ARDS.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

1. To assess the safety of administering cord blood derived mesenchymal stem cell (CB-MSC) infusions for treatment of moderate, severe or critical pneumonia.

SECONDARY OBJECTIVES:

1. In the group of participants who present intubated on ventilator support, assess the proportion that are able to be successfully extubated.
2. In the group of participants who present requiring supplemental oxygen but otherwise breathing without assistance, assess the rate of progression to intubation.
3. Estimate the survival rate at day 30 post treatment separately by group.
4. Determine the treatment effect on clinical parameters, oxygenation and respiratory parameters:

   * Resolution of fever
   * Changes in oxygen demand (increased oxygen saturation at similar FiO2 or decreased FiO2 requirement)
   * Progression to mechanical ventilation
   * Length of Mechanical ventilation
   * Decrease in PEEP in intubated participants
   * Decrease in FiO2 in intubated participants
5. Determine the treatment effect on laboratory markers:

   * Complete blood count
   * CRP
   * Ferritin
   * D Dimer
   * Procalcitonin
   * Cytokine levels
6. Estimate hospitalization and ICU stay.
7. Report on study related adverse events.

OUTLINE:

Currently not shipping cells outside of MD Anderson Cancer Center in Houston.

PILOT STUDY: Patients receive MSCs intravenously (IV) over 1-2 hours on day 1. participants may receive a second infusion of MSCs within 7 days after the first infusion per physician discretion.

PHASE II STUDY: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive MSCs IV over 1-2 hours on day 1. Patients may receive a second infusion of MSCs within 7 days after the first infusion per physician discretion.

ARM II: Patients receive standard of care.

After completion of study treatment, patients are followed up at days 7, 14, 30, 60, and months 6 and 12.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal 18 years.
2. Participants with chest x-ray findings concerning for pneumonia from any cause, with clinical signs suggestive of at least moderate illness such as respiratory rate >20 breaths per minute or with oxygen saturation less than 93% on room air**
3. Participants with COVID-19 associated pneumonia must meet baseline categorization of Moderate, Severe or Critical COVID-19 per FDA Guidance for Industry COVID-19: Developing Drugs and Biologics Products for Treatment or Prevention, February 2021.
4. Negative pregnancy test in a woman with childbearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization.
5. Participant or legally authorized representative consent. Participants with diminished mental capacity may be allowed on to enroll on the study.
6. Because of the nature of COVID-19, participants enrolled on this study with COVID-19 associated pneumonia may have been previously enrolled in other IND trials for their cancer diagnosis or for COVID-19. These enrollments will not exclude them from enrollment to this study.

Exclusion Criteria:

* Moribund participants not expected to survive up to 48 hours
* Participants with severe chronic liver disease (Childs-Pugh score > 10)
* Pregnant and/or lactating women
* Participants on extracorporeal membrane oxygenation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-07-29 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of composite serious adverse events (Phase I) | Within 30 days of the first mesenchymal stem cell (MSC) infusion
  Serious adverse events with be comprised of grade 3 or 4 graft versus host disease or death and will be estimated and reported overall and by group, along with 95% confidence intervals.
Patients alive without grade 3, 4 infusional toxicity (Phase II) | At day 30 post MSC infusion
Patients alive with grade 3 or 4 infusional toxicity (Phase II) | At day 30 post MSC infusion
Patients not alive (Phase II) | At day 30 post MSC infusion

SECONDARY OUTCOMES:
Proportion of successfully extubated patients who present intubated on ventilator support (Phase I) | Up to day 30 post MSC infusion
  Will be estimated and reported with 95% confidence intervals.
Rate of successful progression to intubation in patients who require supplemental oxygen but who are otherwise able to breathe without assistance (Phase I) | Up to day 30 post MSC infusion
  Will be estimated and reported with 95% confidence intervals.
Overall survival rate (Phase I) | At day 30 post MSC infusion
  Will be estimated and reported with 95% confidence intervals.
Survival rate in patients who present intubated on ventilator support (Phase I) | At day 30 post MSC infusion
  Will be estimated and reported with 95% confidence intervals.
Survival rate in patients who require supplemental oxygen but who are otherwise able to breathe without assistance (Phase I) | At day 30 post MSC infusion
  Will be estimated and reported with 95% confidence intervals.
Clinical parameters (Phase I) | Up to day 30 post MSC infusion
  The effect of MSCs on clinical parameters will be assessed. Continuous clinical parameters will be summarized by means, medians, standard deviations, ranges, and quartiles. Categorical parameters will be summarized by frequency tables.
Oxygenation parameters (Phase I) | Up to day 30 post MSC infusion
  The effect of MSCs on oxygenation parameters will be assessed. Continuous oxygenation parameters will be summarized by means, medians, standard deviations, ranges, and quartiles. Categorical parameters will be summarized by frequency tables.
Respiratory parameters (Phase I) | Up to day 30 post MSC infusion
  The effect of MSCs on respiratory parameters will be assessed. Continuous respiratory parameters will be summarized by means, medians, standard deviations, ranges, and quartiles. Categorical parameters will be summarized by frequency tables.
Laboratory markers (Phase I) | Up to day 30 post MSC infusion
  The effect of MSCs on laboratory markers will be assessed. Continuous laboratory parameters will be summarized by means, medians, standard deviations, ranges, and quartiles. Categorical parameters will be summarized by frequency tables.
Hospitalization stay (Phase I) | Up to day 30 post MSC infusion
Intensive care unit stay (Phase I) | Up to day 30 post MSC infusion
Incidence of infusion-related adverse events (Phase I) | Up to day 30 post MSC infusion
  All grades of infusion-related adverse events will be summarized by grade and type.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Olson, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org